CLINICAL TRIAL: NCT02290886
Title: A Multicenter Phase I/II Clinical Trial, Randomized, Controlled With Placebo, Triple Blind to Evaluate Safety, and Indications of Efficiency of the Intravenous Administration of the Therapy With 3 Doses of MSC in Patients With ASL Moderated to Severe
Brief Title: A Multicenter Phase I/II Clinical Trial to Evaluate Safety of Mesenchymal Stem Cell in Patients With Amyotrophic Sclerosis Lateral
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CeTMAd/ELA/2011
Record Dates: First submitted 2014-10-09; First posted 2014-11-14 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: safety evaluation; intravenous administration; 3 doses of autologous MSC; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Intravenous administration of placebo
  Interventions: Other: Intravenous administration of placebo
- 1 million of MSC (Experimental): Intravenous administration of 1 million of MSC/ kg
  Interventions: Drug: Intravenous administration of 1 million of MSC
- 2 million of MSC (Experimental): Intravenous administration of 2 million of MSC/ kg
  Interventions: Drug: Intravenous administration of 2 million of MSC
- 4 million of MSC (Experimental): Intravenous administration of 4 million of MSC/ kg
  Interventions: Drug: Intravenous administration of 4 million of MSC

INTERVENTIONS:
Other: Intravenous administration of placebo
  Arms: Placebo
Drug: Intravenous administration of 1 million of MSC
  Arms: 1 million of MSC
Drug: Intravenous administration of 2 million of MSC
  Arms: 2 million of MSC
Drug: Intravenous administration of 4 million of MSC
  Arms: 4 million of MSC

SUMMARY:
A multicenter phase I/II Clinical trial,randomized, controlled with placebo, triple blind to evaluate the safety of the intravenous administration of 3 doses of autologous mesenchymal stem cells cells from adipose tissue in patients with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
A multicenter phase I/II Clinical trial,randomized, controlled with placebo, triple blind to evaluate the safety of the intravenous administration of 3 doses of autologous mesenchymal stem cells cells from adipose tissue in patients with Amyotrophic Lateral Sclerosis (ALS).

40 patients will be enrolled and will be randomized into one of the following 4 arms:

* 10 patients in the control group (placebo)
* 10 patients received a dose of 1 million MSC / kg
* 10 patients received a dose of 2 million MSC / kg.
* 10 patients received a dose of 4 million MSC / kg

The follow-up phase of each patient from the cell infusion/placebo will be 6 months.

At the time that each patient completed the follow-up period (i.e., 6 months after the infusion of the cellular product or placebo), the blind will be open, and patients who have been assigned to the control group, will receive the cell product as secondary treatment. These patients will be randomized to receive each of the doses used in the first phase. From this point, they begin a second period of follow up of 6 months.

In addition, after 6 months of MSC infusion, every patient will continue in an open extension study for 36 months to assess the safety of MSC.

ELIGIBILITY:
Inclusion Criteria:

1. Women and males over 18-year-old.
2. Good understanding of the protocol and aptitude to grant the informed assent.
3. Diagnosis of sporadic ALS, with diagnosis of certainty, that is to say, definite or probable, in agreement with the criteria of "El Escorial", of the World Federation of Neurology.
4. Forced vital capacity of at least 50 % of the one that would correspond to them for sex, height and age.
5. More than 6 and less than 36 months of evolution of the disease (from the beginning of the symptoms).
6. Possibility of obtaining, at least, 50gr of adipose tissue.
7. Treatment with riluzole, for at least, a month before the inclusion.

Exclusion Criteria:

1. Any concomitant disease that under investigator's criteria could concern the measures of the clinical variables of the trial (hepatic, renal or cardiac insufficiency, diabetes mellitus, etc).
2. Previous therapy with stem cells.
3. Participation in another clinical trial during 3 months previous to the entry in this trial.
4. Any disease lymphoproliferative
5. Tracheostomy and /or gastrostomy.
6. Haemophilia, diathesis hemorrhagic or anticoagulative current therapy.
7. Hypersensitivity known to the bovine foetal whey or the gentamicin.
8. Medical precedents of infection of the HIV or any serious condition of immunocompromised.
9. Positive HBV or HCV serology
10. Levels of creatinine in whey > 3.0 in subjects not submitted to haemodialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Number of adverse serious unexpected reactions or not, attributable to the treatment (SUSSARs or SAE) | 6 months
  To evaluate the safety of the intravenous administration of 3 doses of autologous mesenchymal stem cells (MSC) from adipose tissue in patients with Amyotrophic lateral Sclerosis (ALS) ABSENCE of: complications in the place of the infusion, appearance of a new neurological effect not attributable to the natural progression of this pathology and adverse serious unexpected reactions or not, attributable to the treatment (SUSSARs or SAE)
Complications in the place of the infusion | 6 months
  To evaluate the safety of the intravenous administration of 3 doses of autologous
Appearance of a new neurological effect not attributable to the natural progression of this pathology | 6 months
  To evaluate the safety of the intravenous administration of 3 doses of autologous

SECONDARY OUTCOMES:
Changes in the progression of the disease (modifications in the scale of functionality of the ALS) | 6 months
Changes in the degree of muscular force | 6 months
Changes in the vital forced capacity | 6 months
Changes of the muscular mass estimated by Nuclear Magnetic Resonance (NMR) of the upper and low extremities | 6 months
Changes in neurophysiological parameters and of quality of life | 6 months
Need and time to tracheotomy or permanent assisted ventilation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Óscar Fernández, MD, Study Chair — Hospital Regional U. de Málaga
Locations (4):
- Spain (4):
  - Hospital Regional Universitario Reina Sofía, Córdoba
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen Macarena, Servicio de Neurología, Seville
  - Hospital Universitario Virgen del Rocío, Seville

REFERENCES:
- [Derived] Ilieva H, Maragakis NJ. Motoneuron Disease: Clinical. Adv Neurobiol. 2017;15:191-210. doi: 10.1007/978-3-319-57193-5_7. PMID 28674982